CLINICAL TRIAL: NCT02170038
Title: Open Label, One-way Crossover Study to Assess the in Vivo Formation of Ethinylestradiol Following Single Intramuscular Administration of 200 mg Norethisterone Enantate Compared to Ethinylestradiol Pharmacokinetics After Multiple Doses of a Combined Oral Contraceptive Containing Ethinylestradiol and Levonorgestrel in Healthy Premenopausal Women
Brief Title: Clinical Study Investigating the Conversion of the Contraceptive Compound Norethisterone Within the Body Towards the Contraceptive Compound Ethinylestradiol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17004; 2013-005280-89 (EudraCT Number)
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Pharmacokinetics
Keywords: Drug Kinetics
MeSH Terms: interventions — ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Healthy premenopausal subjects will receive multiple oral doses of Microgynon for 21days
  Interventions: Drug: Microgynon
- Arm 2 (Experimental): Healthy premenopausal subjects will receive a single intramuscular dose of Noristerat
  Interventions: Drug: Noristerat(BAY86-6308)

INTERVENTIONS:
Drug: Microgynon — Subjects will receive 21 daily oral doses of Microgynon tablets containing 0.15 mg levonorgestrel und 0.03 mg ethinylestradiol.
  Arms: Arm 1
Drug: Noristerat(BAY86-6308) — Subjects will receive one intramuscular dose of Noristerat (oily solution for intramuscular injection) containing 200 mg norethisterone enantate.
  Arms: Arm 2

SUMMARY:
The clinical phase I study aims at investigating the conversion of the contraceptive compound norethisterone within the body towards the contraceptive compound ethinylestradiol. Therefore concentrations of ethinylestradiol will be measured from blood samples after administration of a single intramuscular dose of norethisterone. In a comparison arm concentrations of ethinylestradiol will be measured from blood samples after administration of a pill containing ethinylestradiol itself.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subject
* Age: 18 to 45 years (inclusive) at the first screening examination / visit
* Body mass index (BMI): above or equal 18 and below or equal 30 kg / m²
* At least 3 months since delivery, abortion, or lactation before the first screening examination / visit

Exclusion Criteria:

* - Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Liver diseases, kidney diseases, metabolic disorders, thyroid disorders and known or suspected malignant or benign tumors
* Presence or a history of venous or arterial thrombotic/thromboembolic events
* Migraine with neurologic symptoms (complicated migraine)
* Clinically significant depression
* Pancreatitis or a history thereof if associated with severe hypertriglyceridemia
* Use of systemic or topical medicines or substances which oppose the study objectives or which might influence them

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum observed drug concentration of ethinylestradiol at steady state after multiple administrations of Microgynon (Cmax)ss | At different time points on day 21
Area under the concentration-time curve of ethinylestradiol at steady state after multiple administrations of Microgynon {AUC(0-24)}ss | At different time points on day 21
Maximum observed drug concentration of ethinylestradiol after single administration of Noristerat (Cmax) | At different time points upto 8 weeks
Area under the concentration-time curve of ethinylestradiol after single administration of Noristerat (AUC) | At different time points up to 8 weeks
Maximum observed drug concentration of Norethisterone after single administration of Noristerat (Cmax) | At different time points up to 8 weeks
Area under the concentration-time curve of Norethisterone after single administration of Noristerat (AUC) | At different time points up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany